CLINICAL TRIAL: NCT05099575
Title: Different Protocols for Prevention of Atonic Postpartum Hemorrhage During Cesarean Delivery in High Risk Group
Brief Title: Protocols for Prevention of PPH During CS in High Risk Group
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa Wanees Ahmed, Randa Wanees Ahmed, Assiut University
Other Study IDs: Atonic PPH in high risk group
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Atonic PPH
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant women who receive oxytocin
  Interventions: Drug: Syntocinon, papal, misotac
- Pregnant Women who receive carbetocin
  Interventions: Drug: Syntocinon, papal, misotac
- Pregnant women who receive misoprostol
  Interventions: Drug: Syntocinon, papal, misotac
- Pregnant women who receive ergometrine
  Interventions: Drug: Syntocinon, papal, misotac

INTERVENTIONS:
Drug: Syntocinon, papal, misotac — Using different drugs to prevent atonic PPH during CD in high risk group

SUMMARY:
PPH is one of the most leading causes of maternal mortality,. It means loss of 500 ml blood after vaginal delivery and 1000 ml blood after cesarean delivery. Although it's preventable it represents about 27%of maternal deaths. Atony is the main cause of PPH. 70%of PPH corresponds to uterine atony. Uterotonics like oxytocin, misoprostol, ergometrine, carbetocin and combinations of these drugs can be used but until now there is no agreement on medication that can be the most effective.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pregnant full term>37 w 2. Maternal age 19- 40 3.physical state 1&2 4.patient willing to enter the study

Exclusion Criteria:

* 1.who refuse to participate in study 2.immunocomprmized and patients who had contraindicated from any of drugs used 3.patients with hypersensitivity to any drug

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prevention of atonic PPH during CD in high risk group
Sampling Method: Non-Probability Sample
Enrollment: 448 (Estimated)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss | 1 year
  Decrease amount of blood loss

SECONDARY OUTCOMES:
Finding the drug most effective with least adverse effects | 1 year